CLINICAL TRIAL: NCT06009445
Title: Renal Resistive Index by Renal Doppler Ultrasound as a Predictor of Acute Kidney Injury and Evaluation of Fluid Administration in Sepsis Patients: Cohort Study
Brief Title: Renal Resistive Index as a Predictor of Acute Kidney Injury and Evaluation of Fluid Administration in Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Safinaz Abdelkhalek Aboelfetoh, Resident of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Other Study IDs: 36264MS189/5/23
Record Dates: First submitted 2023-08-19; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Renal Resistive Index; Acute Kidney Injury; Sepsis
MeSH Terms: conditions — Acute Kidney Injury; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AKI group: Acute kidney injury (AKI) was defined according to the Kidney Disease Improving Global Outcome (KDIGO) classification using both creatinine and urine output criteria.
  The KDIGO guidelines define AKI as follows:
  * Increase in serum creatinine by ≥0.3 mg/dL (≥26.5 micromol/L) within 48 hours, or
  * Increase in serum creatinine to ≥1.5 times baseline, which is known or presumed to have occurred within the prior seven days, or
  * Urine volume <0.5 mL/kg/hour for six hours
  Interventions: Diagnostic Test: Renal resistive index
- Non AKI group: Patients who will no develop Acute kidney injury (AKI).
  Interventions: Diagnostic Test: Renal resistive index

INTERVENTIONS:
Diagnostic Test: Renal resistive index — The calculation formula for Renal resistive index (RRI) as follows :
  (systolic peak flow velocity _ diastolic minimum flow velocity )/systolic peak flow velocity .
  will be measured with ultrasound-Doppler using an abdominal curvilinear probe ultrasonography by two independent, trained sonographers (who will not be involved in patient care. After visualizing the kidney in ultrasound mode and checking for renal abnormalities, an arcuate or interlobar artery will be localized and three successive doppler measurements at different positions in the kidney (high, middle and low) will be performed, 3 times in each kidney. So a total number of 9 RRI values will be obtained in each kidney.
  The median value of each section will be used and the 3 median values of each kidney will be averaged.
  Other Names: Renal Doppler Ultrasound

SUMMARY:
We aim from this study to investigate the role of renal resistance index (RRI) in evaluation of Acute kidney injury development and fluid administration in sepsis patients considering the change in RRI values over 7 days from admission as a predictor of AKI development

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is one of the most common problems in critically ill patients in the clinic. AKI can be caused by various factors, such as hypovolemia, shock, major surgery, trauma, and heart failure, of which sepsis is the most common

ELIGIBILITY:
Inclusion Criteria:

* Age over 21 years
* meet Sepsis 3 criteria (potential source of infection , host response and organ dysfunction) but not in septic shock.

Exclusion Criteria:

* patients during pregnancy.
* patients with hepatorenal syndrome.
* Poor abdominal echogenicity eg.(morbid obesity ,increase intra abdominal pressure )
* Severe acute or chronic renal insufficiency .
* Dialysis dependency.
* Renal transplantation.
* Known renal artery stenosis.
* Mono-kidney, kidney tumor, anatomic kidney abnormalities.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Tanta university surgical intensive care unit (SICU)
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Prediction of AKI development by renal resistance index (RRI) | 7 days from admission
  AKI was defined according to the Kidney Disease Improving Global Outcome (KDIGO) classification using both creatinine and urine output criteria.
  The KDIGO guidelines define AKI as follows
  * Increase in serum creatinine by ≥0.3 mg/dL (≥26.5 micromol/L) within 48 hours, or
  * Increase in serum creatinine to ≥1.5 times baseline, which is known or presumed to have occurred within the prior seven days, or
  * Urine volume <0.5 mL/kg/hour for six hours

SECONDARY OUTCOMES:
Evaluation of fluid administration | 7 days from admission
  RRI and other hypoperfusion markers after fluid challenge and divided into responder to fluid (Time 1 F) and non responder with noradrenaline administration (Time 1 N) .
Length of ICU stay | 2 months from admission till discharge
  Length of ICU stay till discharge will be measured.
cumulative fluid balance over 7 days | 7 days from admission
  Cumulative fluid balance over 7 days and urine output (intake -output) will be measured.
The incidence of 28 day mortality | 28 days from admission
  The incidence of mortality will be measured at 28 day.

CONTACTS AND LOCATIONS:
Overall Officials: Safinaz A Aboelfetoh, MBBCh, Principal Investigator — Anesthesiology, Faculty of Medicine, Tanta University, Egypt.
Locations (1):
- Tanta University Hospitals, Tanta, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available after the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.